CLINICAL TRIAL: NCT03792490
Title: Inhibition of Rho Kinase (ROCK) With Fasudil as Disease-modifying Treatment for ALS
Acronym: ROCK-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Paul Lingor, International Coordinator, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01742; 2017-003676-31 (EudraCT Number); 01GM1704A (Other Grant/Funding Number: BMBF); 01GM1704B (Other Grant/Funding Number: BMBF); 00013948 (Registry Identifier: DRKS)
Record Dates: First submitted 2018-12-28; First posted 2019-01-03 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Motor neuron disease; Neurodegenerative disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Neurodegenerative Diseases | interventions — fasudil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasudil 30 mg (Experimental): Fasudil (Fasudil hydrochloride hydrate IV solution) Dosage form: intravenous, application over 45 minutes Dosage: 30 mg/ day Frequency: 2 x 15 mg Duration of treatment: 20 days
  Interventions: Drug: Fasudil
- Fasudil 60 mg (Experimental): Fasudil (Fasudil hydrochloride hydrate IV solution) Dosage form: intravenous, application over 45 minutes Dosage: 60 mg/ day Frequency: 2 x 30 mg Duration of treatment: 20 days
  Interventions: Drug: Fasudil
- Placebo (Placebo Comparator): Sodium chloride (NaCl) 0.9% Dosage form: intravenous, application over 45 minutes Dosage: 100 ml Frequency: 2 x Duration of treatment: 20 days Do2 x 1 ml, NaCl 0.9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fasudil — Fasudil hydrochloride hydrate IV solution
  Arms: Fasudil 30 mg; Fasudil 60 mg
Drug: Placebo — Placebo to Fasudil hydrochloride hydrate, NaCl 0,9%
  Arms: Placebo

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disorder and therapeutic options are limited. The rho kinase (ROCK) inhibitor Fasudil was shown to be neuroprotective, induced axonal regeneration and improved survival and behavioral outcome in models of ALS and other neurodegenerative diseases. The aim of this phase IIa, multi-center and double-blind study is to analyze the safety, tolerability and efficacy of fasudil in two different doses compared to placebo in approximately 16 trial sites in Germany, France and Switzerland. Intravenous application of fasudil will be performed in 80 patients and placebo in 40 patients two times daily for 20 treatment days. The hypothesis is that fasudil is safe and well-tolerated and its application will significantly improve the clinical outcome in patients with ALS.

ELIGIBILITY:
Inclusion Criteria:

* Probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria
* Disease duration more than 6 months and less than 24 months (inclusive). Disease onset defined as date of first muscle weakness, excluding fasciculations and cramps
* Vital capacity more than 65% of normal (slow vital capacity; best of three measurements)
* Age: ≥ 18 years
* Patients have to be treated with Riluzole (2 x 50mg/d), must be stable for at least four weeks before randomization
* Patients who have started on Edaravone therapy shall continue Edaravone treatment. Edaravone treatment must not be discontinued for reasons of trial participation.
* Women of childbearing age must be non-lactating and surgically sterile or using a highly effective method of birth control and have a negative pregnancy test. Acceptable methods of birth control with a low failure rate i.e. less than 1% per year) when used consistently and correct are such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner
* Capable of thoroughly understanding all information given and giving full informed consent according to good clinical practice (GCP)
* Patients have to have a valid health insurance, when recruited in a center in France

Exclusion Criteria:

* Previous participation in another clinical study involving trial medication within the preceding 12 weeks or five terminal half times of the longest to be eliminated trial medications (whichever is longer) or previous participation in this trial
* Tracheostomy or continuous assisted ventilation of any type during the preceding three months before randomization or a significant pulmonary disorder not attributed to ALS, which may complicate the evaluation of respiratory function, intermittent non-invasive ventilation is permitted,
* Patients with a history of intracranial bleeding, known intracerebral aneurysms or Moyamoya disease, or positive family history for the above. If only family history positive, magnetic resonance (MR)- or x-ray-based cranial imaging not older than 24 months must confirm absence of bleeding, aneurysms or Moyamoya.
* Gastrostomy
* Any medical condition known to have an association with motor neuron dysfunction or involving neuromuscular weakness or another neurodegenerative disease, e.g. Parkinson's disease (PD) or Alzheimer's disease (AD), which might confound or obscure the diagnosis of ALS
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* Patients with known arterial hypotension (resting blood pressure <90/60 mmHg) or previous hypotensive episodes or requiring treatment for increasing of blood pressure, such as fludrocortisone, midodrine, etilefrine, cafedrine or theodrenaline
* Patients with an uncontrollable or unstable arterial hypertensive disease (resting blood pressure >180 mmHg systolic and/or >120 mmHg diastolic under current antihypertensive medication)
* Known pulmonary hypertension and any medication prescribed for treatment of pulmonary hypertension
* Confirmed hepatic insufficiency or abnormal liver function (stable aspartate transaminase (ASAT) and/or alanine aminotransferase (ALAT) greater than 3 times the upper limit of the normal range) and determined to be non-transient through repeat testing
* Renal insufficiency with a glomerular filtration rate (GFR) <60 ml/min/1,73m² (calculated by Modification of Diet in Renal Disease (MDRD) equation) and determined to be non-transient through repeat testing
* Major psychiatric disorder, significant cognitive impairment or clinically evident dementia precluding evaluation of symptoms
* Hypersensitivity to any component of the study drug
* Liable to be not cooperative or comply with the trial requirements (as assessed by the investigator), or unable to be reached in the case of emergency
* Pregnant or breast-feeding females or females with childbearing potential, if no adequate contraceptive measures are used
* Prisoners or subjects who are involuntary incarcerated
* Patients subject to legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Safety (proportion of patients without treatment-related serious adverse events (SAE) up to day 180) and tolerability (proportion of patients without significant drug intolerance during the treatment period) | From baseline (day 1) to last follow-up (day 180 ± 5)
  Primary endpoint is the proportion of patients without significant drug intolerance during the treatment period (tolerability) and the proportion of patients without treatment-related serious adverse events (SAE) up to day 180 (safety).

SECONDARY OUTCOMES:
Survival time | From baseline (day 1) to end of treatment (day 26 to 30), second follow-up (day 90 ± 4), last follow-up (day 180 ± 5)
ALS Functional Rating Scale (ALSFRS-R) | From baseline (day 1) to end of treatment (day 26 to 30), second follow-up (day 90 ± 4), last follow-up (day 180 ± 5)
  Amyotrophic lateral sclerosis functional rating scale - revised (ALSFRS-R):
  a scale to determine different aspects of functionality in patients with ALS, minimum 0 points, maximum 48 points, derived from a questionnaire with 12 questions, each of which can yield up to 4 points, higher score indicates better functionality
ALS Assessment Questionnaire (ALSAQ-5) | From baseline (day 1) to end of treatment (day 26 to 30), second follow-up (day 90 ± 4), last follow-up (day 180 ± 5)
  Amyotrophic lateral sclerosis assessment questionnaire (ALSAQ-5):
  a patient self-report five-item scale to determine the health status and quality of life in patients with ALS, higher scores show worse quality of life
Edinburgh Cognitive and Behavioral ALS Screen (ECAS) | From baseline (day 1) to end of treatment (day 26 to 30), second follow-up (day 90 ± 4), last follow-up (day 180 ± 5)
  Edinburgh Cognitive and Behavioral Amyotrophic Lateral Sclerosis Screen (ECAS):
  a scale to determine the cognitive function of patients with ALS, minimum 0 points, maximum 136 points, higher scores show better cognitive performance
Motor Unit Number Index (MUNIX) | From baseline (day 1) to end of treatment (day 26 to 30), second follow-up (day 90 ± 4), last follow-up (day 180 ± 5)
  Motor Unit Number Index (MUNIX):
  a neurophysiological method based on surface EMG recordings to estimate the number of motor units, higher scores indicate a higher number of motor units
slow Vital capacity (VC) | From baseline (day 1) to end of treatment (day 26 to 30), second follow-up (day 90 ± 4), last follow-up (day 180 ± 5)
Safety (proportion of patients without treatment-related serious adverse events (SAE) up to end of treatment (day 26 to 30)) and tolerability (proportion of patients without significant drug intolerance during the treatment period) | From baseline (day 1) to end of treatment (day 26 to 30)

CONTACTS AND LOCATIONS:
Locations (15):
- France (4):
  - Centre Hospitalier Universitaire Marseille, Marseille
  - Centre Hospitalier Universitaire Montpellier, Montpellier
  - Centre Hospitalier Universitaire Nice, Nice
  - Centre Hospitalier Universitaire Tours, Tours
- Germany (10):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - University Medical Center Göttingen, Göttingen
  - Universitätsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Ulm, Ulm
  - University of Würzburg, Würzburg
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lingor P, Weber M, Camu W, Friede T, Hilgers R, Leha A, Neuwirth C, Gunther R, Benatar M, Kuzma-Kozakiewicz M, Bidner H, Blankenstein C, Frontini R, Ludolph A, Koch JC; ROCK-ALS Investigators. ROCK-ALS: Protocol for a Randomized, Placebo-Controlled, Double-Blind Phase IIa Trial of Safety, Tolerability and Efficacy of the Rho Kinase (ROCK) Inhibitor Fasudil in Amyotrophic Lateral Sclerosis. Front Neurol. 2019 Mar 27;10:293. doi: 10.3389/fneur.2019.00293. eCollection 2019. PMID 30972018
- [Derived] Koch JC, Leha A, Bidner H, Cordts I, Dorst J, Gunther R, Zeller D, Braun N, Metelmann M, Corcia P, De La Cruz E, Weydt P, Meyer T, Grosskreutz J, Soriani MH, Attarian S, Weishaupt JH, Weyen U, Kuttler J, Zurek G, Rogers ML, Feneberg E, Deschauer M, Neuwirth C, Wuu J, Ludolph AC, Schmidt J, Remane Y, Camu W, Friede T, Benatar M, Weber M, Lingor P; ROCK-ALS Study group. Safety, tolerability, and efficacy of fasudil in amyotrophic lateral sclerosis (ROCK-ALS): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2024 Nov;23(11):1133-1146. doi: 10.1016/S1474-4422(24)00373-9. PMID 39424560
- [Derived] Lingor P, Koch JC, Statland JM, Hussain S, Hennecke C, Wuu J, Langbein T, Ahmed R, Gunther R, Ilse B, Kassubek J, Kollewe K, Kuttler J, Leha A, Lengenfeld T, Meyer T, Neuwirth C, Tostmann R, Benatar M. Challenges and opportunities for Multi-National Investigator-Initiated clinical trials for ALS: European and United States collaborations. Amyotroph Lateral Scler Frontotemporal Degener. 2021 Aug;22(5-6):419-425. doi: 10.1080/21678421.2021.1879866. Epub 2021 Feb 3. PMID 33533663
- See also: Information for patients and physicians — http://rock-als.uni-goettingen.de